CLINICAL TRIAL: NCT02059824
Title: Normal Eyelid Sensation Distribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00051285
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2015-01

CONDITIONS: Normal Eyelid Sensation Distribution
Keywords: Eyelid sensation, aesthesiometer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyelid (Experimental): The selection of the laterality of the eyelid will be randomized
  Interventions: Device: Aesthesiometer

INTERVENTIONS:
Device: Aesthesiometer — The eyelid sensation will be tested on every third by applying the tip of the aesthesiometer filament perpendicular to the eyelid skin and tarsal plate until the filament bent slightly. The filament length will be set at 6 cm (longest length) and applied to the test site 3 times. This process will be repeated 3 times and if the patient verbally responded to the 3rd touch, the number 6 will be recorder.
  If the patient responded less than 3 of the 3 times, the filament will be shortened by 0.5 cm and the test will be repeated. This process will be continued by shortening the filament 0.5 cm each time, until the patient feels the filament touch 3 of 3 times. This filament length number will be recorded as the touch reading for that time period.

SUMMARY:
The purpose of this study is to determine normal eyelid sensation distribution using a Cochet-Bonett Aesthesiometer.

DETAILED DESCRIPTION:
After proper taken consent patients without previous eyelid surgery in the Oculoplastic clinic at Duke Eye Center and Duke Aesthetic Center will be enrolled to test the eyelid sensation distribution using the Cochet-Bonnet aesthesiometer. The aesthesiometer (Luneau ophthalmologie) with a 0.12mm diameter filament was chosen for its ease of use, sensitivity, and safety. This instrument contains a 6 cm long, retractable, flexible monofilament. For any given length, when applied perpendicularly to test surface, the filament will exert a precise pressure before visibly bending. The filament length inversely corresponds to the pressure exerted by the aesthesiometer.

Selection of eyelid laterality will be randomized on the same day of the study. Ipsilateral upper and lower eyelids will be divided in thirds (medial, central and lateral borders) including the margin (fig.2). The eyelid sensation will be tested on every third by applying the tip of the aesthesiometer filament perpendicular to the eyelid skin and tarsal plate until the filament bent slightly. The filament length will be set at 6 cm (longest length) and applied to the test site 3 times. This process will be repeated 3 times and if the patient verbally responded to the 3rd touch, the number 6 will be recorder.

If the patient responded less than 3 of the 3 times, the filament will be shortened by 0.5 cm and the test will be repeated. This process will be continued by shortening the filament 0.5 cm each time, until the patient feels the filament touch 3 of 3 times. This filament length number will be recorded as the touch reading for that time period.

The mean touch thresholds for the various test sites will be compared using a Freidman two-way analysis variant (ANOVA).

ELIGIBILITY:
Inclusion Criteria

* Capable and willing to provide consent
* Has been seen for the first time in the Oculoplastic clinic and does not have previous eyelid surgery
* At least 18 years of age

Exclusion Criteria:

* Unable or unwilling to give consent
* Under 18 years of age
* Previous eyelid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Eyelids' sensation distribution | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Richard, MD, Principal Investigator — Duke Medical Center
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

REFERENCES:
- [Background] McGowan DP, Lawrenson JG, Ruskell GL. Touch sensitivity of the eyelid margin and palpebral conjunctiva. Acta Ophthalmol (Copenh). 1994 Feb;72(1):57-60. doi: 10.1111/j.1755-3768.1994.tb02738.x. PMID 8017198
- [Background] Lowther GE, Hill RM. Sensitivity threshold of the lower lid margin in the course of adaptation to contact lenses. Am J Optom Arch Am Acad Optom. 1968 Sep;45(9):587-94. doi: 10.1097/00006324-196809000-00003. No abstract available. PMID 5245726
- [Background] Black EH, Gladstone GJ, Nesi FA. Eyelid sensation after supratarsal lid crease incision. Ophthalmic Plast Reconstr Surg. 2002 Jan;18(1):45-9. doi: 10.1097/00002341-200201000-00007. PMID 11910324
- [Background] Komiyama O, Wang K, Svensson P, Arendt-Nielsen L, Kawara M, De Laat A. Ethnic differences regarding sensory, pain, and reflex responses in the trigeminal region. Clin Neurophysiol. 2009 Feb;120(2):384-9. doi: 10.1016/j.clinph.2008.11.010. Epub 2008 Dec 24. PMID 19110468
- [Background] Costas PD, Heatley G, Seckel BR. Normal sensation of the human face and neck. Plast Reconstr Surg. 1994 May;93(6):1141-5. doi: 10.1097/00006534-199405000-00005. PMID 8171132